CLINICAL TRIAL: NCT01454934
Title: A Randomized, Open-label, Multicenter, Phase 3 Study to Compare the Efficacy and Safety of Eribulin With Treatment of Physician's Choice in Subjects With Advanced Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E7389-G000-302
Record Dates: First submitted 2011-10-13; First posted 2011-10-19 (Estimated); Results first posted 2017-03-01 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2017-08

CONDITIONS: Non-Small Cell Lung Cancer (NSCLC)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — eribulin; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A (Experimental)
  Interventions: Drug: Eribulin
- Arm B (Active Comparator)
  Interventions: Drug: TPC -Vinorelbine,Gemcitabine,Docetaxel, and Pemetrexed

INTERVENTIONS:
Drug: Eribulin — Administration of eribulin mesylate at a dose of 1.4 mg/m2 i.v. over 2 to 5 minutes on Days 1 and Day 8 of every cycle, where the duration of each cycle is 21 days.
  Arms: Arm A
Drug: TPC -Vinorelbine,Gemcitabine,Docetaxel, and Pemetrexed — * Vinorelbine 30 mg/m2 i.v. on Day 1, every 7 days
  * Gemcitabine 1250 mg/m2 i.v. on Days 1 and 8, every 21 days
  * Docetaxel 75 mg/m2 i.v. on Day 1 every 21 days
  * Pemetrexed 500 mg/m2 i.v. on Day 1 every 21 days (nonsquamous histology only).
  Arms: Arm B

SUMMARY:
This is a randomized, open-label, multicenter, Phase 3 study, comparing efficacy and safety of eribulin with TPC in subjects with advanced and disease progression following at least two prior regimens for advanced disease, which should have included a platinum-based regimen.

ELIGIBILITY:
Inclusion:

Subjects must meet all of the following criteria to be included in this study:

1. Histologically or cytologically confirmed diagnosis of NSCLC.
2. Documented evidence of advanced NSCLC not amenable to surgery or radiotherapy.
3. Confirmation of the presence or absence of EGFR mutations prior to study enrolment in all subjects.
4. Subjects must have received at least two prior regimens for advanced NSCLC, which should have included a platinum-based regimen and, in all subjects with tumors harbouring EGFR mutations, an EGFR TKI.
5. Radiographic evidence of disease progression on, or after, the last anti-cancer regimen prior to study entry.
6. Presence of measurable disease.
7. ECOG performance status of 0, 1, or 2.
8. Adequate bone marrow
9. Adequate renal function.
10. Adequate liver function.
11. Female subjects of child-bearing potential must agree to use two forms of highly effective contraception.
12. Male subjects and their female partners who are of child-bearing potential must agree to use two forms of highly effective contraception.
13. Voluntary agreement to provide written informed consent and the willingness and ability to comply with all aspects of the protocol.
14. Males or females aged at least 18 years (or any age greater than 18 years as determined by country legislation) at the time of informed consent.

Exclusion:

Subjects who meet any of the following criteria will be excluded from this study:

1. Subjects who have received any anti-cancer therapy within 14 days, or five half-lives of the drug (whichever is longer), prior to randomization.
2. Subjects who have not recovered from toxicities as a result of prior anti-cancer therapy to less than Grade 2.
3. Subjects who have previously been treated, or participated in a study with eribulin, whether treated with eribulin or not. The TPC option must not include the same agent which the subject received in a prior regimen.
4. Peripheral neuropathy more than CTCAE Grade 2.
5. Significant cardiovascular impairment.
6. Subjects with a high probability of Long QT Syndrome, or QTc interval >500 ms.
7. Subjects with brain or subdural metastases are not eligible, unless the metastases are asymptomatic and do not require treatment or have been adequately treated by local therapy.
8. Any serious concomitant illness.
9. Known HIV positive, or have an infection requiring treatment.
10. Any malignancy that required treatment, or has shown evidence of recurrence (except for NSCLC, non-melanoma skin cancer, or histologically confirmed complete excision of carcinoma in-situ) during the 5 years prior to study entry.
11. Female subjects must not be pregnant, and must not be breastfeeding.
12. Hypersensitivity to either HalB or HalB chemical derivatives or both, or to any of the excipients of the eribulin formulation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 540 (Actual)
Dates: Start 2011-12-09 (Actual); Primary Completion 2014-05-30 (Actual); Study Completion 2016-05-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (83):
- United States (13):
  - Los Angeles, California
  - Pleasant Hill, California
  - San Diego, California
  - Aurora, Colorado
  - Washington D.C., District of Columbia
  - Port Saint Lucie, Florida
  - Decatur, Illinois
  - Southfield, Michigan
  - Lebanon, New Hampshire
  - Lake Success, New York
  - Portland, Oregon
  - Spokane, Washington
  - Madison, Wisconsin
- Australia (2):
  - Herston, Queensland
  - Frankston, Victoria
- France (12):
  - Strasbourg, Bas Rhin
  - Marseille, Bouches-du-Rhone
  - Marseille, Bouches-duRhone
  - Bordeaux, Gironde
  - Toulouse, Haute Garonne
  - Limoges, Haute Vienne
  - Rennes, Ille Et Vilaine
  - Saint-Herblain, Loire Atlantique
  - Lille, Nord
  - Paris, Paris
  - Pierre-Bénite, Rhone
  - Villejuif, Val De Marne
- Germany (8):
  - Aschaffenburg, Bavaria
  - Gauting, Bavaria
  - Munich, Bavaria
  - Cologne, North Rhine-Westphalia
  - Essen, North Rhine-Westphalia
  - Recklinghausen, North Rhine-Westphalia
  - Mainz, Rhineland-Palatinate
  - Halle, Saxony-Anhalt
- Hong Kong, Hong Kong
- Italy (6):
  - Lido di Camaiore, Lucca
  - Monza, Milano
  - Aviano, Pordenone
  - Cremona
  - Milan
  - Siena
- Japan (18):
  - Nagoya, Aichi-ken
  - Kashiwa-shi, Chiba
  - Fukuoka, Fukuoka
  - Hiroshima, Hiroshima
  - Sapporo, Hokkaido
  - Kobe, Hygo-Ken
  - Akashi-shi, Hyōgo
  - Sendai, Miyagi
  - Nigata-shi, Nigata-Ken
  - Kurashiki-shi, Okayama-ken
  - Habinko-shi, Osaka
  - Osaka, Osaka
  - Osakasayama-shi, Osaka
  - Sunto-gun, Shizuoka
  - Chūōku, Tokyo-to
  - Kōtoku, Tokyo-To
  - Ube-shi, Yamaguchi
  - Kitaadachi-gun
- Poland (5):
  - Gdansk
  - Mrozy
  - Otwock
  - Sczedin
  - Warsazawa
- Russia (3):
  - Barnaul
  - Novosibirsk
  - Saint Petersburg
- Singapore, Singapore
- South Korea (3):
  - Seongnam-si, Gyeonggi-do
  - Suwon, Gyeonggi-do
  - Seoul, Korea
- Spain (5):
  - Sabadell, Barcelona
  - Terrassa, Barcelona
  - Pamplona, Navarre
  - Barcelona
  - Madrid
- Taiwan (3):
  - Taichung
  - Tainan
  - Taipei
- United Kingdom (3):
  - London, Greater London
  - Manchester, Greater Manchester
  - Sutton, Surrey

REFERENCES:
- [Derived] Katakami N, Felip E, Spigel DR, Kim JH, Olivo M, Guo M, Nokihara H, Yang JC, Iannotti N, Satouchi M, Barlesi F. A randomized, open-label, multicenter, phase 3 study to compare the efficacy and safety of eribulin to treatment of physician's choice in patients with advanced non-small cell lung cancer. Ann Oncol. 2017 Sep 1;28(9):2241-2247. doi: 10.1093/annonc/mdx284. PMID 28911085

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 735 participants were screened. Of these, 195 screen failed due to failure to meet inclusion/exclusion criteria, adverse events, withdrawal of consent, or other reason and were not randomized into the study. A total of 540 participants were randomized into the study. Of these, 3 were discontinued prior to treatment.
Groups:
- Arm A: Eribulin Mesylate: Eribulin mesylate (1.4 milligram per square meter [mg/m^2]) was administered intravenously (IV) over 2 to 5 minutes on Day 1 and Day 8 of every cycle, where the duration of each cycle is 21 days.
- Arm B: Vinorelbine, Gemcitabine, Docetaxel, or Pemetrexed: Treatment of Physician's Choice (TPC): Vinorelbine (30 mg/m^2) was administered IV on Day 1 every 7 days, Gemcitabine (1250 mg/m^2) was administered IV on Days 1 and 8 every 21 days (or 1000 mg/m^2 IV on Days 1, 8, and 15 every 28 days), Docetaxel (75 mg/m^2) was administered IV on Day 1 every 21 days, or Pemetrexed (500 mg/m^2) was administered IV on Day 1 every 21 days (nonsquamous histology only).
Period: Overall Study
Arm/Group | Arm A: Eribulin Mesylate | Arm B: Vinorelbine, Gemcitabine, Docetaxel, or Pemetrexed
Started | 270 | 270
Completed | 0 | 0
Not Completed | 270 | 270
Not completed — Clinical progression | 28 | 25
Not completed — Other | 6 | 17
Not completed — Adverse Event | 28 | 24
Not completed — Withdrawn consent | 2 | 5
Not completed — Withdrawal by Subject | 11 | 15
Not completed — Disease progression | 194 | 181
Not completed — Lost to Follow-up | 0 | 1
Not completed — Not treated | 1 | 2

BASELINE CHARACTERISTICS:
Population: Full analysis set included all randomized participants.
Groups:
- Arm A: Eribulin Mesylate: Eribulin mesylate (1.4 mg/m^2) was administered IV over 2 to 5 minutes on Day 1 and Day 8 of every cycle, where the duration of each cycle is 21 days.
- Arm B: Vinorelbine, Gemcitabine, Docetaxel, or Pemetrexed: TPC: Vinorelbine (30 mg/m^2) was administered IV on Day 1 every 7 days, Gemcitabine (1250 mg/m^2) was administered IV on Days 1 and 8 every 21 days (or 1000 mg/m^2 IV on Days 1, 8, and 15 every 28 days), Docetaxel (75 mg/m^2) was administered IV on Day 1 every 21 days, or Pemetrexed (500 mg/m^2) was administered IV on Day 1 every 21 days (nonsquamous histology only).
- Total: Total of all reporting groups
Arm/Group | Arm A: Eribulin Mesylate | Arm B: Vinorelbine, Gemcitabine, Docetaxel, or Pemetrexed | Total
Number analyzed (Participants) | 270 | 270 | 540
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.4 (9.62) | 60.8 (9.32) | 61.1 (9.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 107 | 101 | 208
  Male | 163 | 169 | 332

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: The OS was defined as the time in months from the date of randomization to the date of death, regardless of cause. In the absence of confirmation of death, the participants were censored either at the date that participant was last known to be alive or the date of study cut-off, whichever was earlier. The two treatment arms were compared using the log-rank test, stratified by histology, TPC option, and geographic region; and the treatment difference between eribulin mesylate and TPC was tested at a significance level of 0.05 (2-sided). Kaplan-Meier (K-M) survival probabilities for each arm were plotted over time. The treatment effect was estimated by fitting a Cox Proportional Hazards model to the OS times including treatment arm as a factor and histology, TPC option and geographic region as strata.
Time Frame: Randomization (Day 1) until date of death from any cause, or 37 months
Population: Full analysis set included all randomized participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A: Eribulin Mesylate | Arm B: Vinorelbine, Gemcitabine, Docetaxel, or Pemetrexed
Number analyzed (Participants) | 270 | 270
months | 9.5 [7.4 to 11.4] | 9.5 [8.5 to 11.3]
Statistical Analysis 1: Comparison: Arm A: Eribulin Mesylate vs Arm B: Vinorelbine, Gemcitabine, Docetaxel, or Pemetrexed; OS was compared between eribulin and TPC testing the following null hypothesis: H0: OS in Arm A (eribulin) is equal to OS in Arm B (TPC) against the alternative: H1: OS in Arm A (eribulin) is not equal to OS in Arm B (TPC); Test type: Superiority or Other; p = 0.1343, Log Rank — P-value was calculated from a 2-sided long-rank test stratified by histology, TPC option, and geographic region; Hazard Ratio (HR) = 1.16, 95% CI 2-sided [0.95 to 1.41] — Hazard Ratio was based on a Cox regression model including treatment as covariate, and histology, TPC option and geographic region as strata

2. Secondary Outcome: Progression Free Survival (PFS) by Response Evaluation Criteria in Solid Tumors (RECIST)
Description: PFS was defined as the time from the date of randomization to the date of first documentation of disease progression, or date of death, whichever occurred first. The difference in PFS (based on the tumor response evaluation as determined by the investigator) between eribulin mesylate and TPC was evaluated using the log rank test, stratified by histology, TPC option, and geographic region, tested at an alpha level of 0.05 (2-sided). PFS censoring rules will be defined in the SAP and follow Federal Department of Agriculture (FDA) guidance.
Time Frame: Randomization (Day 1) until date of disease progression or death (whichever occurred first), or 37 months
Population: Full analysis set included all randomized participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A: Eribulin Mesylate | Arm B: Vinorelbine, Gemcitabine, Docetaxel, or Pemetrexed
Number analyzed (Participants) | 270 | 270
months | 3.0 [2.6 to 3.9] | 2.8 [2.6 to 3.6]
Statistical Analysis 1: Comparison: Arm A: Eribulin Mesylate vs Arm B: Vinorelbine, Gemcitabine, Docetaxel, or Pemetrexed; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.3946, Log Rank — P-value was calculated from a 2-sided long-rank test stratified by histology, TPC option, and geographic region; Hazard Ratio (HR) = 1.09, 95% CI 2-sided [0.90 to 1.32] — The hazard ratio was based on a Cox regression model including treatment as covariate, and histology, TPC option, and geographic region as strata

3. Secondary Outcome: Objective Response Rate (ORR)
Description: The ORR was defined as the proportion of participants with best overall response of complete response (CR) or partial response (PR) per RECIST criteria. The ORR was estimated by study arm based on the tumor response evaluation as determined by the investigator, according to RECIST 1.1. Participants with unknown response were treated as non-responders. The statistical difference in ORR between treatment arms was evaluated using the Cochran-Mantel-Haenszel (CMH) chi-square test with histology, TPC option, and geographic region as strata, tested at an alpha level of 0.05 (2-sided). The 95 percent confidence interval (CI) was calculated using Clopper Pearson method.
Time Frame: Randomization (Day 1) to CR or PR
Population: Full analysis set included all randomized participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A: Eribulin Mesylate | Arm B: Vinorelbine, Gemcitabine, Docetaxel, or Pemetrexed
Number analyzed (Participants) | 270 | 270
percentage of participants | 12.2 [8.6 to 16.7] | 15.2 [11.1 to 20.0]
Statistical Analysis 1: Comparison: Arm A: Eribulin Mesylate vs Arm B: Vinorelbine, Gemcitabine, Docetaxel, or Pemetrexed; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.3034, Cochran-Mantel-Haenszel — The P-value was stratified by histology, TPC option, and geographic region

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (AEs) and serious adverse events (SAEs) were collected from the first dose of study treatment to thirty days after final dose of study medication. Participants were followed for approximately 37 months.
Description: Safety analysis set included all randomized participants who received at least one dose of study treatment. AEs were graded on a 5-point scale according to Common Terminology for Adverse Events (CTCAE) version 4.0. All AEs graded 4 or 5 were considered serious.
Arm/Group | Arm A: Eribulin Mesylate | Arm B: Vinorelbine, Gemcitabine, Docetaxel, or Pemetrexed
All-Cause Mortality (participants affected / at risk) | 28/269 | 21/268
Serious Adverse Events (participants affected / at risk) | 96/269 | 86/268
Other Adverse Events (participants affected / at risk) | 254/269 | 261/268
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: Eribulin Mesylate (N=269) | Arm B: Vinorelbine, Gemcitabine, Docetaxel, or Pemetrexed (N=268)
Anaemia (Blood and lymphatic system disorders) | 2 | 2
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 3 | 7
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 1
Neutropenia (Blood and lymphatic system disorders) | 4 | 3
Acute coronary syndrome (Cardiac disorders) | 0 | 1
Angina unstable (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 1
Cardiac failure (Cardiac disorders) | 1 | 0
Coronary artery thrombosis (Cardiac disorders) | 1 | 0
Myocardial ischaemia (Cardiac disorders) | 2 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 2
Constipation (Gastrointestinal disorders) | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Large intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1
Oesophageal stenosis (Gastrointestinal disorders) | 0 | 1
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 1 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Asthenia (General disorders) | 2 | 3
Chest pain (General disorders) | 0 | 1
Device failure (General disorders) | 0 | 1
Face oedema (General disorders) | 0 | 1
Fatigue (General disorders) | 0 | 3
General physical health deterioration (General disorders) | 13 | 12
Non-cardiac chest pain (General disorders) | 2 | 1
Pain (General disorders) | 1 | 0
Pyrexia (General disorders) | 3 | 3
Hepatic cirrhosis (Hepatobiliary disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 0 | 1
Bronchitis (Infections and infestations) | 0 | 2
Bronchopneumonia (Infections and infestations) | 1 | 1
Cellulitis (Infections and infestations) | 1 | 0
Escherichia sepsis (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 1 | 0
Lung abscess (Infections and infestations) | 0 | 1
Lung infection (Infections and infestations) | 2 | 1
Neutropenic sepsis (Infections and infestations) | 2 | 2
Oral candidiasis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 12 | 5
Pseudomembranous colitis (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 2 | 3
Sepsis (Infections and infestations) | 1 | 2
Septic shock (Infections and infestations) | 1 | 0
Staphylococcal sepsis (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0
Wound infection fungal (Infections and infestations) | 1 | 0
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Ilium fracture (Injury, poisoning and procedural complications) | 1 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 | 0
Blood phosphorus decreased (Investigations) | 0 | 1
Neutrophil count decreased (Investigations) | 1 | 2
White blood cell count decreased (Investigations) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 3
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 4 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Polydipsia (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 4
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastatic pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Brain oedema (Nervous system disorders) | 1 | 0
Cerebral infarction (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 1
Coma (Nervous system disorders) | 0 | 1
Seizure (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1
Embolic cerebral infarction (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 0
Monoplegia (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 2 | 0
Fear (Psychiatric disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9 | 10
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 6
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Deep vein thrombosis (Vascular disorders) | 1 | 1
Hypotension (Vascular disorders) | 0 | 1
Jugular vein thrombosis (Vascular disorders) | 1 | 2
Superior vena cava syndrome (Vascular disorders) | 0 | 2
Superior vena cava stenosis (Vascular disorders) | 1 | 0
Venous thrombosis limb (Vascular disorders) | 1 | 0
Hydrocephalus (Nervous system disorders) | 0 | 1
Cataract (Eye disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: Eribulin Mesylate (N=269) | Arm B: Vinorelbine, Gemcitabine, Docetaxel, or Pemetrexed (N=268)
Anaemia (Blood and lymphatic system disorders) | 59 | 72
Leukopenia (Blood and lymphatic system disorders) | 27 | 28
Neutropenia (Blood and lymphatic system disorders) | 92 | 74
Abdominal Pain (Gastrointestinal disorders) | 13 | 19
Abdominal Pain Upper (Gastrointestinal disorders) | 17 | 17
Constipation (Gastrointestinal disorders) | 63 | 63
Diarrhoea (Gastrointestinal disorders) | 38 | 45
Nausea (Gastrointestinal disorders) | 73 | 78
Stomatitis (Gastrointestinal disorders) | 43 | 34
Vomiting (Gastrointestinal disorders) | 29 | 38
Asthenia (General disorders) | 59 | 56
Fatigue (General disorders) | 66 | 62
Malaise (General disorders) | 22 | 29
Oedema peripheral (General disorders) | 40 | 31
Pyrexia (General disorders) | 47 | 50
Upper respiratory tract infection (Infections and infestations) | 13 | 14
Alanine aminotransferase increased (Investigations) | 19 | 23
Aspartate aminotransferase increased (Investigations) | 17 | 17
Neutrophil count decreased (Investigations) | 60 | 58
Weight decreased (Investigations) | 20 | 15
White blood cell count decreased (Investigations) | 55 | 57
Decreased appetite (Metabolism and nutrition disorders) | 98 | 68
Arthralgia (Musculoskeletal and connective tissue disorders) | 15 | 18
Back pain (Musculoskeletal and connective tissue disorders) | 24 | 21
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 14 | 7
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 14 | 9
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 19 | 24
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 22 | 14
Myalgia (Musculoskeletal and connective tissue disorders) | 28 | 26
Pain in extremity (Musculoskeletal and connective tissue disorders) | 13 | 14
Dizziness (Nervous system disorders) | 14 | 19
Dysgeusia (Nervous system disorders) | 25 | 16
Headache (Nervous system disorders) | 35 | 21
Paraesthesia (Nervous system disorders) | 21 | 6
Peripheral sensory neuropathy (Nervous system disorders) | 44 | 24
Insomnia (Psychiatric disorders) | 16 | 20
Cough (Respiratory, thoracic and mediastinal disorders) | 42 | 42
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 57 | 52
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 19 | 20
Productive cough (Respiratory, thoracic and mediastinal disorders) | 16 | 14
Alopecia (Skin and subcutaneous tissue disorders) | 81 | 42
Rash (Skin and subcutaneous tissue disorders) | 17 | 24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No